CLINICAL TRIAL: NCT06952556
Title: A Randomized, Single-blind, Single-center Study Measuring the Effects of Adductor Canal Block Combined With IPACK Infiltration Compared to Adductor Canal Block Alone on Post-operative Pain and Opioid Consumption in Patients Undergoing HTO/DFO/TTO
Brief Title: Adductor Canal Block and IPACK Block vs. Isolated Adductor Canal Block for Post-Operative Analgesia Following HTO/DFO/TTO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-01855
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adductor Canal Block (ACB) + IPACK Block (Experimental): Participants receive ACB with IPACK block.
  Interventions: Drug: ACB; Drug: IPACK block
- Isolated Adductor Canal Block (Active Comparator): Participants receive ACB only.
  Interventions: Drug: ACB

INTERVENTIONS:
Drug: ACB — 15 mL of 0.25% Bupivacaine block of the saphenous nerve injected under ultrasound guidance via adductor canal.
Drug: IPACK block — IPACK block with 20 mL of 0.25% Bupivacaine injected into the Interspace between the Popliteal Artery and Capsule of the Knee
  Arms: Adductor Canal Block (ACB) + IPACK Block

SUMMARY:
A randomized, single-blind, single-center study measuring the effects of adductor canal block combined with IPACK infiltration compared to adductor canal block alone on post-operative pain and opioid consumption in patients undergoing high tibial osteotomy (HTO)/distal femoral osteotomy (DFO)/tibial tubercle osteotomy (TTO).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age
* Patients undergoing HTO/DFO/TTO.
* American Society of Anesthesiologists (ASA) I or II

Exclusion Criteria:

* Patients younger than 18 and older than 75.
* Patients with multi-ligament injury
* Patients undergoing concomitant cartilage procedure or ACLR.
* Patients with a history of chronic pain that have used opioids for pain management for 3 months or longer.
* Patients who are allergic to oxycodone;
* Patients with diagnosed or self-reported cognitive dysfunction;
* Patients with a history of neurologic disorder that can interfere with pain sensation;
* Patients with a history of drug or recorded alcohol abuse;
* Patients who are unable to understand or follow instructions;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
* Patients with an allergy or contraindication to any of the medications used in the study, or patients with a contraindication to any study procedures;
* Patients with a BMI over 45;
* Any patient that the investigators feel cannot comply with all study related procedures;
* Any pregnant patient; assessed via urine pregnancy test in the preoperative area as part of standard preoperative surgical protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Opioid Utilization for First 24 Hours Post-Surgery | Up to Hour 24 Post-Procedure (Post-Operative Day 1 [POD 1])
  Opioid utilization for the first 24 hours after surgery, including during surgery, calculated as oral morphine equivalent.

SECONDARY OUTCOMES:
Length of Stay in PACU | Post-Operation (POD 0 - typically up to 3 hours)
  Length of time the patient is in the PACU prior to discharge.
Patient-Reported Visual Analogue Scale (VAS) Score - Baseline | Baseline
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score in Post-Anesthesia Care Unit (PACU) | Post-Operation (POD 0 - typically up to 3 hours)
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score - Post-Operative Day 1 (POD 1) | POD 1
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score - Post-Operative Day 2 (POD 2) | POD 2
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score - Post-Operative Day 3 (POD 3) | POD 3
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score - Post-Operative Day 7 (POD 7) | POD 7
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Patient-Reported VAS Score - Month 6 Follow-Up | Month 6 Post-Operation
  Patients rate their pain score on a scale from 0 to 10 (0 being no pain and 10 being the worst imaginable pain); the total score is the response.
Knee injury and Osteoarthritis Outcome Score (KOOS) - Physical Function Shortform (KOOS-PS) Score - Baseline | Baseline
  7-item assessment of how well participants are able to perform different activities. Each item is rated on a 5-point Likert scale (0 to 4), with 0 representing "none" and 4 representing "extreme". The raw score is the sum of responses and is converted to a total score ranging from 0-100, where higher scores indicate greater function.
KOOS-PS Score - Month 6 Follow-Up | Month 6 Post-Operation
  7-item assessment of how well participants are able to perform different activities. Each item is rated on a 5-point Likert scale (0 to 4), with 0 representing "none" and 4 representing "extreme". The raw score is the sum of responses and is converted to a total score ranging from 0-100, where higher scores indicate greater function.
Kujala Score / Anterior Knee Pain Scale (AKPS) - Baseline | Baseline
  13-item self-report questionnaire that assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. The total score is the sum of responses and ranges from 0 to 100, with 100 being the highest possible score. Lower scores reflect greater pain and disability.
Kujala Score / AKPS - Month 6 Follow-Up | Month 6 Post-Operation
  13-item self-report questionnaire that assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. The total score is the sum of responses and ranges from 0 to 100, with 100 being the highest possible score. Lower scores reflect greater pain and disability.
Tegner Activity Scale (TAS) Score - Baseline | Baseline
  The Tegner Activity Scale (TAS) is a 1-item, self-administered questionnaire used to assess a patient's ability to engage in work and sports activities. The item is rated on a scale of 0 to 10, with 0 representing maximum disability and 10 representing elite sports participation. The total score is the item response.
Tegner Activity Scale (TAS) Score - Month 6 Follow-Up | Month 6 Post-Operation
  The Tegner Activity Scale (TAS) is a 1-item, self-administered questionnaire used to assess a patient's ability to engage in work and sports activities. The item is rated on a scale of 0 to 10, with 0 representing maximum disability and 10 representing elite sports participation. The total score is the item response.

CONTACTS AND LOCATIONS:
Overall Officials: Laith Jazrawi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The Investigators will not be sharing this information with other researchers beyond publishing our findings in a scientific journal.